CLINICAL TRIAL: NCT00721877
Title: Clinical Study of Resveratrol on Drug and Carcinogen Metabolizing Enzymes
Brief Title: Resveratrol in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2009-00895; NCI-2009-00895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07-0376-04; BIO07-054; CDR0000656389; 07-0376-04 (Other: Arizona Cancer Center - Tucson); UAZ06-8-01 (Other: DCP); P30CA023074 (NIH); N01CN35158 (NIH)
Record Dates: First submitted 2008-07-24; First posted 2008-07-25 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2013-03

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — Resveratrol

ARMS (1):
- Arm I (Experimental): Participants receive oral resveratrol once daily for 4 weeks.
  Interventions: Drug: resveratrol; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: resveratrol — Given orally
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Resveratrol may prevent cancer in healthy people. Studying samples of blood and urine in the laboratory from participants who are taking resveratrol may help doctors learn more about how this drug is used by the body. This phase I trial is studying the side effects of resveratrol and to see how it works in healthy adult participants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of resveratrol on human cytochrome P450 (CYP) enzyme activity in healthy adult participants.

SECONDARY OBJECTIVES:

I. To determine the modulation effect on phase II detoxification enzymes. II. To evaluate safety in participants treated with this drug.

OUTLINE:

Participants receive oral resveratrol once daily for 4 weeks.

Patients complete a daily diary documenting adverse events and an intake calendar for recording the daily intake of any non-routine medications.

Participants undergo blood sample collection periodically. Lymphocytes are isolated and analyzed for baseline GST activity and level. Serum is analyzed to determine bilirubin levels to be used as surrogate UGT 1A1 activity. Analyses of CYP probe drugs will be performed using high performance liquid chromatography (HPLC) assays. A sensitive ELISA assay will be used for quantitative analyses. Urine samples are collected periodically and drug and metabolite levels will be analyzed.

After completion of study treatment, participants are followed for 2 weeks.

ELIGIBILITY:
Criteria:

* Healthy adult participants meeting the following criteria:
* Limit cruciferous vegetables to no more than one serving each week for about 6 weeks
* Limit resveratrol-containing foods (i.e., wine, peanuts, mulberries, grapes, cranberries, blueberries, and huckleberries) to no more than one serving each per day for about 6 weeks
* No caffeine-containing food or beverages (e.g., coffee, colas, chocolate, or over-the-counter medications) or food items that have been reported to affect drug/carcinogen metabolizing enzymes (e.g., grapefruit, grapefruit juice, cruciferous vegetables, and food cooked over charcoal) beginning 72 hours before and until 8 hours after each set of CYP probe drug administration
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelet count >= 100,000/uL
* Total bilirubin =< 2.0 mg/dL
* AST/ALT =< 1.5 times upper limit of normal (ULN)
* Creatinine =< ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must have a resting systolic blood pressure >= 100 mm Hg at screening and prior to probe drug administration
* Must not consume more than three drinks of alcohol per week on average
* No prior invasive cancers (i.e., non-skin cancer) within the past 5 years
* No history of allergic reactions to resveratrol-containing products or CYP probe drugs (e.g, caffeine, dextromethorphan, losartan, or buspirone)
* No uncontrolled intercurrent illness including, but not limited to, any of the following:
* Ongoing or active infection
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Cardiac arrhythmia
* Psychiatric illness or social situation that would limit compliance with study requirements
* No over-the-counter medications beginning 72 hours before and until 8 hours after each CYP probe drug administration
* No participation in another clinical intervention trial within the past 3 months
* No concurrent medications or supplements that are known CYP enzyme inducers or inhibitors
* No concurrent herbal medicines, dietary supplements, or above-standard vitamins or minerals (a standard daily multivitamin or mineral supplement is acceptable)
* Non-smoking, defined as not currently smoking or stopped smoking more than 1 year ago
* Normal liver and renal function
* Able and willing to adhere to the following dietary restrictions:
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Modulation of CYP enzyme activities | From baseline to end of resveratrol intervention
  Will be assessed by a comparison of CYP enzyme activities from baseline to end of resveratrol intervention. CYP1A2, 2D6, 2C9, and 3A4 activity will be assessed by plasma paraxanthine/caffeine ratio, urinary dextromethorphan/dextrophan ratio, urinary losartan/losartan metabolite ratio, and area under the plasma buspirone concentration-time curve, respectively. The primary analysis will consist of paired t-tests of differences in log values from baseline to end of intervention (equivalent to log of the ratio).

SECONDARY OUTCOMES:
Changes in Phase II enzyme activity | From baseline to end of resveratrol intervention
  GST activity and GST-pi level in blood lymphocytes and serum bilirubin levels will be used to assess Phase II enzyme activity. Paired t-tests of differences in values from baseline to end of intervention will be used, with a 2-sided significance level of 0.0167 for the three tests.
Safety evaluation using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 6 weeks
  Any adverse events will be presented descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Hui (Sherry) Chow, Principal Investigator — Arizona Cancer Center - Tucson
Locations (1):
- Arizona Cancer Center - Tucson, Tucson, Arizona, United States